CLINICAL TRIAL: NCT06176027
Title: Therapeutic Effect of Chemotherapy Azacytidine Plus CAOLD Regimen on Patients With Relapsed/Refractory Peripheral T-Cell Lymphomas
Brief Title: Azacytidine Plus CAOLD Regimen in Relapsed/Refractory Peripheral T-Cell Lymphomas
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Navy General Hospital, Beijing (Other)
Collaborators: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Liren Qian, Associate Chief Physician, Associate Professor, Navy General Hospital, Beijing
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NavyGHB-008
Record Dates: First submitted 2023-08-05; First posted 2023-12-19 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Relapsed Peripheral T-Cell Lymphomas; Refractory Peripheral T-Cell Lymphomas
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Azacytidine plus CAOLD regimen (Experimental): Patients were treated by Azacytidine plus CAOLD regimen
  Interventions: Drug: Azacytidine plus CAOLD regimen

INTERVENTIONS:
Drug: Azacytidine plus CAOLD regimen — Patients were treated by Azacytidine(75 mg/m2 on days 1-7) plus CAOLD regimen (cyclophosphamide 400mg/m2 qd d1; cytarabine 30mg/m2 qd d1-d4; vindesine 2mg/m2 qd d1; pegaspargase 2500iu/m2 qd d2; dexamethasone 7.5mg/m2 qd d1-d5)

SUMMARY:
This is a multicenter prospective single arm phase II study. The purpose of this study is to evaluate the safety and efficiency of azacytidine combined with CAOLD Regimen in the treatment of relapsed/refractory peripheral t-cell lymphomas.

DETAILED DESCRIPTION:
The investigators will evaluate response rate, progression free survival (PFS), overall survival (OS), and toxicity of azacytidine combined with CAOLD Regimen in relapsed/refractory peripheral t-cell lymphomas.

ELIGIBILITY:
Inclusion Criteria:

Patients must satisfy all following criteria to be enrolled in the study:

* Pathologically confirmed angioimmunoblastic T-cell lymphoma according World Health Organization (WHO) classification;
* Patient is ≥ 18 years of age at the time of signing the informed consent form (ICF).
* Patient must understand and voluntarily sign an ICF prior to any study-specific assessments/procedures being conducted;
* Patient is willing and able to adhere to the study visit schedule and other protocol requirements;
* Relapsed (after partial or complete response) or refractory AITL after at least one line of systemic therapy (there is no mandatory resting period after the previous treatment as long as the biochemistry and hematology labs meet the inclusion criteria as below.)
* Meet the following lab criteria:

  * Absolute Neutrophil Count (ANC) ≥ 1,5 x 10^9/L (≥ 1 x 10^9/L if bone marrow (BM) involvement by lymphoma)
  * Platelet ≥ 75 x 10^9/L (≥ 50 x 10^9/L if BM involvement by lymphoma)
  * Hemoglobin ≥ 8 g/dL.
* Anticipated life expectancy at least 3 months

Exclusion Criteria:

* Active or uncontrolled infections requiring systemic treatment within 14 days before enrollment;
* Any instability of systemic disease, including but not limited to severe cardiac, liver, kidney, or metabolic disease need therapy;
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2030-09-01 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | 1 year
  ORR was defined as the proportion of patients who achieved CR or PR as their best response

SECONDARY OUTCOMES:
Overall Survival (OS) | through study completion, an average of 2 year
  OS was defined as time from diagnosis to death from any cause or the last follow-up
Progression Free Survival (PFS) | 18 months
  PFS using local assessment of progressive disease according to Lugano Response Criteria (2014)

CONTACTS AND LOCATIONS:
Overall Officials: Liren Qian, PhD, Study Chair — Navy General Hospital, Beijing
Locations (1):
- Navy General Hospital, Beijing, Beijing Municipality, China